CLINICAL TRIAL: NCT05146258
Title: The Effectivity of the Voiding School for Symptom Reduction and Quality of Life in Children With Lower Urinary Tract Symptoms
Brief Title: Voiding Class Study for Symptom Reduction and Quality of Life in Children With LUTS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10501/10502/10504
Record Dates: First submitted 2021-10-19; First posted 2021-12-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Voiding class; Quality of Life; Children
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lower urinary tract dysfunction (LUTD) is a common pathology within children and shows a wide spectrum of lower urinary tract symptoms (LUTS). These symptoms have a significant impact on a child's well-being. For the treatment of LUTS in children urotherapy, a non-medicamentous form of therapy, is implemented as standard therapy. It can be described as a bladder re-education and rehabilitation programme where the participants are informed on the anatomy and physiology of the normal and pathological urinary system. Urotherapy has been offered as individual therapy for a long time but is now also offered as group therapy (the voiding school). This is, as compared to the individual therapy, more cost-effective and gives the participants the feeling not to be alone in the situation. The effectiveness of the individual therapy for children with LUTD has already been determined, however little research has been done on the effectiveness of urotherapy in group (the voiding class). The present study wants to investigate the effect of the group therapy on the symptoms and quality of life of children with LUTD.

DETAILED DESCRIPTION:
The current study is a prospective cohort-study in which information of the impact of the voiding class on the symptoms and well-being of the children is obtained through two questionnaires, respectively the Vancouver Symptom Score for Dysfunctional Elimination Syndrome (VSSDES) and the Paediatric Incontinence Questionnaire (PinQ). Participants of this study are as well asked to complete drinking and voiding charts and nocturnal diaries. These questionnaires and documents are filled in before and after the voiding class. The collected data will be further analysed statistically trough Statistical Package for the Social Sciences (SPPS), to determine significant improvements in symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* children (5-12 years old)
* children with LUTS
* children who follow voiding school, with or without previously failed training

Exclusion Criteria:

* children >12 years ol and <5 years old
* children who suffer from solely faecal problems without lower urinary tract symptoms
* children who are currently following a different kind of therapy concerning the LUTS, than VC
* children with neurological disorders or anatomical variations of the bladder
* children who underwent surgical intervention of the bladder

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Lower Urinary Tract Dysfunctions attending the group urotherapy, the voiding school
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Lower Urinary Tract Symptoms - VVSDES | through study completion, average of 3 months
  Amount of LUTS before and after the voiding class measured by the Vancouver symptom score for dysfunctional elimination syndrome (VSSDES)
Well-being of the child - PinQ | through study completion, average of 3 months
  The effect of the voiding class on the QoL measured by the Paediatric incontinence questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Samijn, dr., Principal Investigator — Ghent University Hospital/Ghent University
Locations (1):
- Ghent University Hospital/Ghent University, Ghent, East Flanders, Belgium